CLINICAL TRIAL: NCT06996938
Title: PrEVE: Evaluation of the Acceptability and Impact of a Sexual Health Screening and Prevention Program for Vulnerable Women in the Greater Paris Region
Brief Title: Evaluation of the Acceptability and Impact of a Sexual Health Screening and Prevention Program for Vulnerable Women
Acronym: PrEVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de Recherches et d'Etude sur la Pathologie Tropicale et le Sida (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CREPATS 18; 2024-A01338-39 (Other: ANSM)
Record Dates: First submitted 2025-01-24; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Vulnerable Population
MeSH Terms: interventions — Seroconversion

STUDY DESIGN:
Intervention Model Description: The PrEVE study is a prospective, community-based study conducted in the Île-de-France region. It assesses the acceptability of a sexual health prevention pathway including screening by rapid diagnostic orientation tests (TROD) HIV, hepatitis and syphilis among women in vulnerable situations, by consulting at a place dedicated to the precarious.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vulnerable women (Experimental): This is a prospective study, designed to evaluate the use of a sexual health prevention pathway including screening by rapid diagnostic orientation tests (TROD) HIV, Hepatitis, syphilis and the use of a sexual health prevention course for women in vulnerable situations (VF) living in the Île-de-France region.
  Interventions: Diagnostic Test: Rapid diagnostic orientation tests (TROD) HIV, Hepatitis, syphilis

INTERVENTIONS:
Diagnostic Test: Rapid diagnostic orientation tests (TROD) HIV, Hepatitis, syphilis — The following information will be collected :
  * Socio-demographic characteristics
  * Lifestyle
  * Health status
  * Access to care and support in care
  * Life events/violence
  Knowledge of HIV prevention will be assessed
  It will be proposed to screen for potentially serious STIs in the absence of specific management. If one of these infections is detected, the women will be referred and accompanied to a specialized consultation in the medical centers participating in the study
  Women's needs in terms of health and access to care will be assessed: infections, gynecology, psychology, management of individual violence, sexual in particular, prophylaxis with regard to HIV

SUMMARY:
Globally, women accounted for more than half of people living with HIV (53%) in 2022. In France, 54% of new infections were heterosexual in 2022, 71% of whom were born abroad, mainly in sub-Saharan Africa (74%). Among women, 80% of new cases were born abroad, of which at least 30% contracted HIV after arriving in France, often in connection with social vulnerability as shown by the French study Parcours. In the Paris region, 1,243 new cases among women were registered between 2018 and 2021 (about 300 per year).

Unstable housing, experiences of violence, lack of residence permits and sex trade increase the risk of HIV among women. Positive test migrants often report a higher frequency of forced sex. These women also face high risks of other STIs, unwanted pregnancies, violence and mental health problems.

PrEP is a means of preventing HIV infection by taking an antiretroviral drug, which has been fully proven to be effective in the form of tablets or injections. Pre-Exposure Prophylaxis (PrEP) is part of a comprehensive prevention service pathway.

Despite the free availability of PrEP in France from 2027 and essential monitoring tools for men and women at high risk, women at risk remain largely uncovered by prevention initiatives, making them a "hidden population" under-studied. In France, recent data show that only 5% of PrEP users are women, compared to 95% of men, mainly men who have sex with men (MSM).

Several factors hinder access to PrEP, including limited knowledge of available services, misperceptions of risk (because women rarely initiate sexual intercourse), fear of stigma and lack of resources. In addition, France lacks comprehensive programs that integrate health care, sexual health, mental health and social and legal support for these women.

The PrEVE study aims to demonstrate that the involvement of community-based organizations can play an important role in engaging and retaining women in vulnerable situations in a sexual health program. This program provides information, screening and prophylaxis to meet the specific sexual health needs of vulnerable women.

DETAILED DESCRIPTION:
Overall, HIV prevalence among girls and women is higher than that of boys and men since the 2000s. For example, UNAIDS data in 2022 shows that 53% of people living with HIV (PLHIV) are girls and women, or about 21 million people, and 46% of new HIV infections are girls and women.

This difference is due to a higher risk of HIV infection among girls and young women, especially in Africa : UNAIDS pointed out in 2018 that HIV infections among girls and young women aged 15-19 are about twice as high globally as among boys and young men of the same age.

In France, women represent about 35% of PLHIV. Data from the French national hospital cohort of HIV infection show that 1,243 women were newly treated between 2018 and 2021 in Ile de France (IDF), which is about 300 new women taken care of per year. If you consider the population from sub-Saharan Africa, it represents 76% of women living with HIV (FVVIH) in IDF.

Women are at greater risk than men of HIV and other sexually transmitted infections (STIs) because of biological, anatomical characteristics that make transmission from male to female easier. Women have a larger mucous membrane area exposed to pathogens and infectious fluids during heterosexual sex and are likely to experience greater tissue damage.

Girls and women often face multiple, interconnected social, cultural and economic inequalities and are at increased risk of acquiring HIV and sexually transmitted infections (STIs).

Globally, girls and women make up the majority of illiterate people (63%) and the poorest people (52% in 2021). In addition, gender inequalities have been amplified by the COVID-19 health crisis that has led to a significant increase in poverty rates among women. Low educational attainment and poor socio-economic status were associated with an increased risk of HIV infection among women.

The COINCIDE study focused on the IDF epidemic, with the objective of mapping new diagnoses of HIV infection between 2014 and 2021. In total, 10,827 newly-supported PLHIV were included, of which 3,327 (31%) were women living with HIV (VVIH), they were 36 years old median, 86% foreign born and almost a third (31%) were diagnosed at an advanced stage of infection (CD4 < 200/mm3 or AIDS). 75% of the FVVIH lived outside Paris (41% in small-crown departments 92, 93, 94 and 34% in Grande Couronne -77, 78, 91, 95) and above all, that at least 30% of them had a precarious housing (homeless or housed by a third party) at the time of taking charge, reflecting the high level of poverty among this population. Foreign-born FVVIH, which make up the vast majority of IDF's FVVIH, had a 16 times higher risk of having precarious housing compared to men who have sex with men (MSM), after adjustment in place of residence, age and immunoclinical stage at diagnosis (COINCIDE study, unpublished data).

Vulnerability is a particular dimension of women's health and is not sufficiently taken into account. There is a strong link between social disconnection, precariousness and health degradation. It was estimated that access to care for men in precarious situations is five times lower than the population average, with a gap nine times smaller for women.

Access to information and prevention in the field of sexual health is less in France among women who are precarious and/or migrants. The majority of young girls and women aged 15-24 in Africa do not have full knowledge about HIV. Lack of information on HIV prevention and the inability to use such information in sexual relations, including in the context of marriage, They undermine women's ability to negotiate condom use and engage in safer sex practices.

Access to information, HIV and STI testing, PrEP (Pre-Exposure Prophylaxis) prevention for women, especially those who are migrants, is very poor. Thus, 4.6% of PrEP recipients in France are women, compared to a majority use to 97% by men, mainly MSM. Moreover, women are less able to negotiate their protection during sexual intercourse by the condom because of their precarious social situation ;

Lack of information means that too many women consider AIDS to be a male disease and are unaware of their vulnerability to the virus ;

In France, the Parcours study showed that 41% of women born in sub-Saharan Africa are infected after their arrival in France due to a socio-economic vulnerability that exposes them in an increased way. The precarious living conditions of these women expose them to sexual violence, to the exchange of sexual relations for shelter, where negotiation of the use of condoms is impossible. Indeed, the difficulties of women born abroad, the family and professional upheavals that accompany their migration to France have a major impact on their mental health and sexuality.

Worldwide, 35% of women have experienced physical and/or sexual violence at some point in their lives. UNICEF reports that at least one in 10 girls is sexually abused before the age of 18. Exposure to childhood violence, especially sexual violence, increases the risk of HIV infection.

According to the Ministry of the Interior, approximately 210,000 cases of domestic violence against women were registered in 2022. Young women aged 25-39 are overrepresented among the victims (about half), while 15% of these victims are foreign-born. These figures would underestimate the real extent of the problem since, according to the Genesis 2021 victimization survey, only one in four victims of domestic violence report their experiences to security services.

In 2021, one woman living in metropolitan France aged 18 to 74 years out of six reported having experienced sexual violence by a partner at least once since the age of 15, most often repeated. 17.8% of these women reported having been sexually abused at least once since the age of 15 by a non-partner In addition to increasing the risk of HIV infection, this violence has many short and long-term adverse consequences on the physical and mental health of victims: increased risk of use of psychoactive substances, increased risk of developing post-traumatic stress disorder (PTSD), sleep disorders, depressive symptoms, and suicidal ideation. In addition, victims of sexual violence have difficulties accessing specific care due to the scarcity of specialized support in health centres.

More generally, the lack of knowledge about the frequency of these forms of violence and their consequences is a hindrance to their management, even within specialized teams. This care must be multidisciplinary, provided by trained professionals and adapted to the individual situation of each woman.

In the general population, women are more affected by mental health disorders such as depressive syndromes and anxiety than men. In 2017, the prevalence of a characterized depressive syndrome was twice as high among women (13.0% vs 6.4%) compared to men in France. This high risk of mental health disorders is partly explained by an increased risk among women to be subjected to gender-based and sexual violence. Violence against women, which includes domestic and sexual violence linked to impaired mental health.

The use of psychotropic drugs among 15-75 year olds in 2010 was twice as high among women (22%) than men (12.9%). This female consumption increases with age: 11.5% for the 15-34 year old ; 23.5% for the 35-54 year old ; 32.6% for the 55-75 year old.

Women in vulnerable and precarious situations, particularly when born abroad, given the heavy toll paid to HIV infection, are a major key population to target for HIV prevention. This also highlights the need for gender-specific approaches to HIV prevention strategies.

Data on barriers and factors facilitating HIV testing in women are scarce in the international literature. The few studies on the subject suggest that perceived risks, fear, knowledge about testing and stigma will be the main barriers to HIV testing among women outside of the country.

Data on knowledge and perceptions of PrEP in women are also scarce. In addition, the adoption of PrEP by women is limited, in France (less than 5% of PrEP users) but also worldwide.

Thus, understanding the individual, contextual and environmental factors that influence PrEP adoption and HIV testing among women at risk of HIV infection is essential to improving targeted interventions.

Ikambere, "the welcoming house" in Kinyarwanda, was founded in 1997 by Bernadette Rwegera to meet the urgent needs of HIV-positive migrant women, often isolated and in great insecurity. The association offers a safe haven and comprehensive support, integrating therapeutic aspects and social integration.

The association also supports women who face serious health problems and live in very precarious economic and social conditions. It is one of the first associations to have integrated health mediators, perceived as essential for establishing a bond of trust, a prerequisite for continued access to care and its long-term follow-up.

In the Ile de France region, where the number of vulnerable women is particularly high and they represent a population at high risk of acquiring and transmitting STI, it is urgent to implement a specialized intervention. However, despite this urgency, the profiles, specific needs and characteristics of vulnerable women (VW) in terms of prevention and care remain largely unknown and understudied. To date, no comprehensive approach in France takes into account the dimensions of physical, sexual and mental health as well astrauma, in addition to the social and legal support necessary for the care of women in vulnerable situations.

It is in this context that the PrEVE study stands out, conducted by specialized community and association actors, it aims to assess the specific needs of vulnerable women in terms of sexual health and support victims of violence, the acceptability and feasibility of a sexual health pathway including STI screening and prevention measures.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 years of age or older
* Living in Ile de France
* In a vulnerable situation with at least one of the following two situations:

  * Social/economic vulnerability (without personal residence or residence permit of less than 2 years or expiring in less than 1 year or without social security/AME/PUMA (ex CMU)
  * Sexual vulnerability: occasional paid sex worker
* Able to understand the objectives of the study
* Having been informed of the study objectives and not opposed to participating in the study.
* Having signed the consent form prior to any examination being performed in the study.

Exclusion Criteria:

• Person protected by law, or not in a position to express their consent or subject to a measure of guardianship or safeguard of justice

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
Number of women in vulnerable situations who accepted sexual health testing the HIV/Syphilis | between Day 0 and Month 6
  Measure HIV/Syphilis assessed by rapid test using INSTI multiplex
Number of women in vulnerable situations who accepted sexual health testing the VHB | between Day 0 and Month 6
  Measure VHB assessed by rapid test using TOYO Ag HBs/ac anti-HBS
Number of women in vulnerable situations who accepted sexual health testing the VHC | between Day 0 and Month 6
  Measure VHC assessed by rapid test using INSTI HCV

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Pitie-Salpetriere Hospital, Paris
  - IKAMBERE Association, Saint-Denis, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No